CLINICAL TRIAL: NCT04859439
Title: An Open-label, Single-dose, Phase I Clinical Study to Assess the Pharmacokinetics and Safety of DBPR108 Tablets in Subjects With Varying Degrees of Renal Impairment Compared to the Control Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of DBPR108 in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-CSP-009
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — DBPR108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mild Renal Impairment (Experimental): Subjects will receive a single dose of 100 mg DBPR108
  Interventions: Drug: DBPR108 tablets
- Moderate Renal Impairment (Experimental): Subjects will receive a single dose of 100 mg DBPR108
  Interventions: Drug: DBPR108 tablets
- Severe Renal function (Experimental): Subjects will receive a single dose of 100 mg DBPR108
  Interventions: Drug: DBPR108 tablets
- Kidney failure (Experimental): Subjects will receive a single dose of 100 mg DBPR108
  Interventions: Drug: DBPR108 tablets
- Normal Renal function (Experimental): Subjects will receive a single dose of 100 mg DBPR108
  Interventions: Drug: DBPR108 tablets

INTERVENTIONS:
Drug: DBPR108 tablets — Drug: DBPR108, tablet, oral
  Other Names: DBPR108

SUMMARY:
This is an open-label, single-dose study to evaluate the pharmacokinetics and safety of DBPR108 in subjects with mild, moderate, severe renal impairment and subjects with kidney failure compared to the matched control subjects with normal renal function.

DETAILED DESCRIPTION:
This is an open-label, single-dose Phase I study that evaluate the pharmacokinetics, safety, and tolerability of a single dose of DBPR108 100 mg in subjects with mild, moderate, and severe renal impairment (RI), subjects with kidney failure and the control subjects with normal renal function. This study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period (Day 1 to Day 3), and a follow-up call on Day 6.

Subjects will be enrolled in the following groups:

Estimated glomerular filtration rate (eGFR) will be calculated based on Modification of Diet in Renal Disease (MDRD) equation at screening.

(A) mild renal impairment (60 ≤ eGFR≤ 89 mL/min/1.73m2); (B) moderate renal impairment (30 ≤ eGFR≤ 59 mL/min/1.73m2); (C) severe renal impairment (15 ≤ eGFR≤ 29 mL/min/1.73m2); (D) kidney failure (<15 mL/min/1.73m2, not on hemodialysis); (E) control subjects with normal renal function will be matched with subjects with HI by weight, age, and sex (eGFR≥90 mL/min/1.73m2).

Approximately 8 subjects will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions；
* 18 years to 79 years (inclusive), male and female；
* Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height2 (m2))；
* Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration；

Subjects with RI only:

* Subjects with medically stable RI corresponding to the Classifications of Renal Function based on eGFR: mild RI: 60 to 89 ml/min/1.73m2; moderate RI: 30 to 59 ml/min/1.73m2, severe RI:15-29 ml/min/1.73m2, kidney failure:<15 ml/min/1.73m2 (not on hemodialysis);
* Not in use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening, except for the medication necessary for RI/ other comorbidities with no effect on the study drug absorption, distribution, metabolism, or excretion (last more than four weeks in good compliance);
* Based on physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests (serum potassium: 3.5-5.5 mmol/L);

Subjects with normal renal function only:

* Weight, age, and sex must be matched with subjects with HI;
* eGFR≥90 ml/min/1.73m2;
* Not in use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening, except for the medication necessary for underlying conditions other than renal disease with no effect on the study drug absorption, distribution, metabolism, or excretion (last more than four weeks in good compliance).

Exclusion Criteria:

All subjects:

* Subjects who have a history of allergic conditions (such as asthma, urticaria), or have a history of allergy to two or more drugs or food, or may be allergic to the test drug and the related compounds;
* Have a history of severe and uncontrolled diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematologic, mental/nervous systems diseases within one year prior to screening；
* Have previously undergone surgery that may affect drug absorption, distribution, metabolism, or excretion (e.g., subtotal gastrectomy), or who have a scheduled surgical plan during the study period;
* Use of any DPP-IV enzyme inhibitor within 2 weeks prior to the screening;
* Drug abuse, or positive urine drug screen at screening；
* Smoking more than 5 cigarettes per day within 3 months prior to screening；
* Average alcohol intake is more than 28g alcohol (male) or 14g (female) per week (14g ≈ 497mL beer, or 44mL spirits with low alcohol content, or 145mL wine) within the 3 months prior to screening, or taking any alcohol within 48 hours before dosing, or a positive ethanol breath test at screening;
* Consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 hours before the administration, or have strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc.；
* Participation in another clinical trial within 3 months before screening；
* Blood donation (or blood loss) ≥400 mL, or receiving whole blood transfusions or erythrocyte suspension transfusions within 3 months prior to the screening；
* Have acute hepatitis or a chronic liver disease; aspartate aminotransferase (AST), alanine aminotransferase (ALT) or bilirubin > 2 × upper limit of normal；
* Have a positive result for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or anti-treponema pallidum specific antibody；
* A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial；
* Currently receiving, or unable to refrain from expected concomitant cytochrome (CYP) 3A inhibitors and inducers;
* Not suitable for this study as judged by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Cmax
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  AUC0-t
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  AUC0-inf
The pharmacokinetic parameters of DBPR108 in urine | predose and 48 hours after dosing
  Ae
The pharmacokinetic parameters of DBPR108 in urine | predose and 48 hours after dosing
  fe
The pharmacokinetic parameters of DBPR108 in urine | predose and 48 hours after dosing
  CLR

SECONDARY OUTCOMES:
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Tmax
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  t1/2
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Vz/F
The pharmacokinetic parameters of DBPR108 in plasma | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  CL/F
The pharmacokinetic parameters of DBPR108 in urine | predose and 48 hours after dosing
  Ae(t1-t2)
The number of volunteers with adverse events as a measure of safety and tolerability | Day 1 to Day 6
  The number of volunteers with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China